CLINICAL TRIAL: NCT05088447
Title: A Study to Investigate Cystic Fibrosis Pulmonary Exacerbations and the Lung Microbiome
Status: Terminated | Type: Observational
Why Stopped: Change in research plan
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 32509
Record Dates: First submitted 2015-05-18; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stable Disease: 15 control "stable disease" participants
- Frequent Exacerbation Cohort: 15 experimental "frequent exacerbation cohort"

SUMMARY:
The present application proposes to study the role the composition of the pediatric CF airway microbiota plays in frequent pulmonary exacerbations in pediatric CF patients.

In order to accomplish this goal the dynamics of the composition of the CF airway microbiota in two distinct subsets of pediatric patients with CF will be characterized, those with frequent pulmonary exacerbations and clinically stable children. Clinical measures of pulmonary function, patient reported symptoms, sleep quality, and antibiotic usage will be recorded, and these findings will be correlated with the lung microbiota data.

This strategy promises to identify the key characteristics of the pediatric CF microbiota, which can in turn be used as noninvasive markers to identify those patients at a higher risk for experiencing repeated pulmonary exacerbations.

DETAILED DESCRIPTION:
Acute pulmonary exacerbations cause significant morbidity in the lives of children with cystic fibrosis (CF). As the etiologies of exacerbations continue to be defined, characterizing the role of the pulmonary microbiota in chronic infection and inflammation provides an opportunity for insight into the pathophysiology of CF.

This point is particularly true for a subset of pediatric CF patients with severe disease and frequent exacerbations.

The present application proposes to test the overall hypothesis that the composition of the pediatric CF airway microbiota plays an etiologic role in frequent pulmonary exacerbations in pediatric CF patients. To address the working hypothesis, next-generation sequencing based 16S rRNA sequencing will be undertaken to dissect the microbiome of pediatric CF patients subject to frequent pulmonary exacerbations, relative to the microbiome in clinically stable CF patients. This strategy promises to more specifically and definitively identify the key characteristics of the pediatric CF microbiota that are associated with the occurrence of exacerbations. Record clinical measures of pulmonary function, patient reported symptoms, sleep quality, and antibiotic usage, and correlate these findings with the lung microbiota data. This insight would in turn provide noninvasive biomarkers to identify those patients at a higher risk for experiencing repeated pulmonary exacerbations, which over the long-term significantly compromise lung function.

ELIGIBILITY:
Pulmonary Exacerbation Cohort

Inclusion Criteria:

1. Diagnosis of CF (: a. One or more clinical features of CF AND (b or c); b. Sweat chloride > 60 mEq/L; c. Two known CF mutations)
2. 3 or more admissions with an admitting diagnosis of pulmonary exacerbation, requiring IV antibiotics, within the 12 month period prior to study enrollment.

Clinically Stable Disease Cohort

Inclusion Criteria:

1. Diagnosis of CF (: a. One or more clinical features of CF AND (b or c); b. Sweat chloride > 60 mEq/L; c. Two known CF mutations)
2. Age and gender matched to Pulmonary Exacerbation Cohort
3. No hospitalizations with an admitting diagnosis of pulmonary exacerbation, within the 12 month period prior to study enrollment.

Exclusion criteria for both groups includes:

1. History of intolerance or inability to tolerate the induced sputum protocol.
2. History of organ transplantation.
3. Any patient that in discretion of the investigators is not suitable.
4. Any clinically unstable participants.

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: For the "Pulmonary Exacerbation Cohort," recruitment will be of cystic fibrosis pediatric patients with 3 or more hospital admissions with an admitting diagnosis of pulmonary exacerbation, requiring IV antibiotics, within the 12 month period prior to study enrollment, irrespective of race or ethnicity.
  This cohort will be matched with a "Clinically Stable Disease Cohort" which is matched by age, gender and CF genotype, irrespective of race or ethnicity.
  Ages recruited will be children, adolescents and young adults with Cystic Fibrosis from age 0-22 years.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in lung microbiome profile | Baseline - 3 years
  Lung microbiome in Cystic Fibrosis pulmonary exacerbations

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tracy, MD, Principal Investigator — Stanford University
Locations (1):
- Cystic Fibrosis Clinic, LPCH, Palo Alto, California, United States